CLINICAL TRIAL: NCT05044676
Title: Assessment of Circulating Immune Cells as a Prognostic Factor in Patients With Advanced Hepatocellular Carcinoma Treated With Immunotherapy
Brief Title: Immune Cells as a New Biomarker of Response in Patients Treated by Immunotherapy for Advanced Hepatocellular Carcinoma
Acronym: IMMUNOCELL
Status: Terminated | Type: Observational
Why Stopped: Abandon of study
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210845
Record Dates: First submitted 2021-07-05; First posted 2021-09-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; immunotherapy; immune cells; biomarkers
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with hepatocellular carcinoma: Patients with an indication for treatment with Atezolizumab / Bevacizumab for the management of an advanced disciplinary hepatocellular carcinoma in a multidisciplinary consultation meeting.
  Interventions: Other: patients with hepatocellular carcinoma

INTERVENTIONS:
Other: patients with hepatocellular carcinoma — The response of the hepatocellular carcinoma to treatment will be evaluated as part of the care

SUMMARY:
Hepatocellular carcinoma (HCC) is the third leading cause of cancer death worldwide. Treatment options for advanced HCC remain very limited. Until recently, multikinase inhibitor were the gold standard for advanced hepatocellular carcinoma but associated with poor outcome and important side effects. Recently, the positive results of the Imbrave 150 study (a randomized study comparing Atezolizumab + Bevacizumab versus Sorafenib) prompted us to redefine our management strategy for advanced hepatocellular carcinoma by proposing the combination of Atezolizumab/Bevacizumab as treatment first-line in patients with advanced hepatocellular carcinoma. However, only 1/3 of the patients will respond to the combination of treatment and identifying predictive factors of response and new immune checkpoint inhibitors in order to target more tumors appear as a major issue. In this context, recent work has underlined the importance of the activating CD226/DNAM-1 receptor as an original immunotherapeutic target in various cancers (solid and hematopoietic tumors). CD226 is a transmembrane receptor that is part of the immunoglobulin superfamily. It is expressed by most T lymphocytes (CD8+, CD4+), by Natural Killer (NK) cells, by promoting their cytotoxicity.

The investigators propose to prospectively analyze the frequency and phenotype (expression of CD226) of circulating immune cells before the initiation of treatment with Atezolizumab/Bevacizumab, 3 weeks after the first injection and its variation to determine whether this biomarker could predict the response to the treatment.

DETAILED DESCRIPTION:
It is now widely accepted that inflammation is an essential element in tumor development. Liver tissue is very sensitive to inflammation and harbors immune system effectors capable of preventing the onset of a chronic inflammatory response. However, in case of chronic liver diseases, chronic inflammation will favor fibrosis progression and tumor development. Hepatocellular carcinoma (HCC) is the third leading cause of cancer death worldwide. Treatment options for advanced HCC remain very limited. Until recently, multikinase inhibitor were the gold standard for advanced hepatocellular carcinoma but associated with poor outcome and important side effects. Recently, immune checkpoint inhibitors, have emerged as an innovative anti-tumor strategy to restore an anti-tumor immune response, as illustrated by recent positive results of immunotherapy in oncology with prolonged responses in some patients. The initial results of immunotherapy in advanced hepatocellular carcinoma as monotherapy have been disappointing. However, combinations of immunotherapy and anti-VEGF antibodies or between immunotherapy and tyrosine kinase inhibitors are currently being tested in order to potentiate the effect of immunotherapy and to obtain higher rates of anti-tumor response. Recently, the positive results of the Imbrave 150 study (a randomized study comparing Atezolizumab + Bevacizumab versus Sorafenib) prompted us to redefine our management strategy for advanced hepatocellular carcinoma by proposing the combination of Atezolizumab/Bevacizumab as treatment first-line in patients with advanced hepatocellular carcinoma. However, only 1/3 of the patients will respond to the combination of treatment and identifying predictive factors of response and new immune checkpoint inhibitors in order to target more tumors appear as a major issue. In this context, recent work has underlined the importance of the activating CD226/DNAM-1 receptor as an original immunotherapeutic target in various cancers (solid and hematopoietic tumors). CD226 is a transmembrane receptor that is part of the immunoglobulin superfamily. It is expressed by most T lymphocytes (CD8+, CD4+), by Natural Killer (NK) cells, by promoting their cytotoxicity. The ligands for CD226 are the molecules CD112 and CD155, which are overexpressed in many tumors and are associated with a poor prognosis for patients. Recent data show that the decrease in CD226 expression on the surface of anti-tumor-containing immune effectors may be associated with resistance to anti-PD1/PDL1 immunotherapies. To date, the involvement of CD226 and its ligands in liver tumorigenesis is completely unknown. The use of Atezolizumab/Bevacizumab in France is a unique opportunity to conduct a pilot study on clinical, biological, histological, molecular and immune prognostic and predictive factors in patients treated with the Atezolizumab/Bevacizumab combination.

The investigators hypothese that a decrease in CD226 expression on the surface of CD8+ T lymphocytes (CTLs) and NK cells before the initiation of treatment with Atezolizumab/Bevacizumab could be associated with decrease response to the treatment and therefore associated with poor outcome of the patient. The investigators propose to prospectively analyze the frequency and phenotype (expression of CD226) of circulating immune cells before the initiation of treatment with Atezolizumab/ Bevacizumab, 3 weeks after the first injection (day of the second infusion) and its variation to determine whether this biomarker could predict the response to the treatment. The investigators will also perform an analysis of the histological and pathology characteristics of the tumor and non-tumor liver of the same patient before the initiation of treatment with Atezolizumab/ Bevacizumab with the ultimate objective of developing a predictive prognostic score for treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Advanced hepatocellular carcinoma with an indication of systemic therapy by Atezolizumab-Bevacizumab
* At least one measurable untreated lesion
* ECOS performance status of 0 or 1

Exclusion Criteria:

* HIV/ immunosuppressive treatment
* Active of history of autoimmune disease or immune deficiency
* Priori history of liver transplantation or systemic porto shunt
* Pregnant of breastfeeding women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for treatment with Atezolizumab / Bevacizumab for the management of an advanced disciplinary hepatocellular carcinoma in a multidisciplinary consultation meeting (RCP).
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Measurement of the frequency expression of CD226 at baseline | at baseline
Measurement of the frequency expression of CD226 3 weeks after the start of treatment | 3 weeks after the start of treatment
Measurement of the phenotype of expression of CD226at baseline | at baseline
Measurement of the phenotype of expression of CD226 3 weeks after the start of treatment | 3 weeks after the start of treatment

SECONDARY OUTCOMES:
Frequency of expression of CD226 to predict Overall survival (OS) | at baseline and 3 weeks after the start of treatment
  Overall survival determined according to death status or not
phenotype expression of CD226 to predict Overall survival (OS) | at baseline and 3 weeks after the start of treatment
  Overall survival determined according to death status or not
Correlation between pathology features (tumoral and non-tumoral liver) and the frequency and phenotype of expression of CD226 | At inclusion
  Comparison of the immune cells (frequency and phenotype) in the blood and liver tissues (tumoral and non-tumoral liver)

CONTACTS AND LOCATIONS:
Overall Officials: Manon ALLAIRE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service hépato-gastroentérologie, Hôpital la Pitié-Salpêtrière, Paris, France, France